CLINICAL TRIAL: NCT00603590
Title: Phase II Study of Heart Polypill in Primary Prevention of Cardiovascular Disease - Safety and Efficacy
Brief Title: Phase II Study of Heart Polypill Safety and Efficacy in Primary Prevention of Cardiovascular Disease
Acronym: Polypill
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: University of Birmingham (Other)
Responsible Party: Reza Malekzadeh, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 301/148; CCT-NAPN 15388
Record Dates: First submitted 2008-01-01; First posted 2008-01-29 (Estimated); Results first posted 2009-06-23 (Estimated); Last update posted 2009-10-02 (Estimated); Status verified 2009-09

CONDITIONS: Cardiovascular Disease; Hypertension; Hyperlipidemia; Heart Disease
Keywords: Cardiovascular disease; primary prevention; Polypill; efficacy; safety; ADR; Diabetes; Adherence; Compliance
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Hyperlipidemias; Heart Diseases; Diabetes Mellitus; Patient Compliance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Polypill (Experimental): Fixed dose combination therapy with Aspirin 81mg, Hydrochlorothiazide 12.5mg, Enalapril 2.5mg and Atorvastatin 20mg
  Interventions: Drug: Polypill
- Control (Placebo Comparator): Identical placebo
  Interventions: Drug: Placebo drug

INTERVENTIONS:
Drug: Polypill — Fixed dose combination therapy - aspirin 81mg, hydrochlorothiazide 12.5mg, enalapril 2.5mg and atorvastatin 20mg Once daily
  Arms: Polypill
Drug: Placebo drug — Inactive tablet Once a day Identical in appearance to intervention drug
  Arms: Control

SUMMARY:
Cardiovascular is a major cause of mortality in Iran, accounting for 45.7% of deaths. In Golestan (North Eastern Iran) preliminary findings from follow-up of the Golestan Cohort are consistent with national figures: with 45% (at least 22 of 48 deaths) of all deaths attributed to cardiovascular events. Cardiovascular diseases will become an increasing problem as the Iranian population ages.

In 2003 Law and Wald proposed prevention of cardiovascular disease using fixed-dose combination therapy combining antihypertensive, lipid lowering and antiplatelet drugs in a single preparation. They proposed that this treatment should be offered to all persons at high risk of cardiovascular disease whether or not they have elevated blood pressure or elevated serum lipid concentrations.

This pilot study aims to investigate the safety and efficacy of fixed-dose combination therapy with two antihypertensive drugs, aspirin and atorvastatin in a population who would not currently be considered eligible for antihypertensive treatment or for lipid lowering treatment.

Methods:

This is a double-blind randomized controlled trial. The intervention group will be assigned to take a tablet consisting of a single daily tablet comprising Aspirin 81mg, Hydrochlorothiazide 12.5mg, Enalapril 2.5mg and Atorvastatin 20mg. The control group will be assigned to an identical placebo.

The population studied includes men aged 50 to 80 (inclusive) and women aged 55 to 80 (inclusive) who are currently not eligible for or taking antihypertensive or lipid lowering therapy. Persons who are found at baseline to have blood pressure >160/100 mm Hg, total cholesterol >240mg/dL, existing cardiovascular disease or to be taking antihypertensive ore lipid lowering therapy are excluded.

It is intended to randomize and follow up 500 subjects for 12 months. The primary outcome for the purpose of sample size calculation is change in systolic blood pressure. Additional outcomes include change in diastolic blood pressure, change in LDL cholesterol and occurrence of adverse events.

ELIGIBILITY:
Inclusion criteria

All men over 50 to 80 and all women 55 to 80 who are resident in Kalaleh, Golestan, for at least one year.

Exclusion criteria

* Existing cardiovascular disease (stroke, transient ischaemic attack, myocardial infarction or angina)
* Already taking antihypertensive drugs, aspirin or statins
* Already have clinical indications for treatment with antihypertensive drugs, aspirin or statins.

  * Blood pressure >160/100 mm Hg
  * Total Cholesterol > 240 mg/dL (or LDL >190 mg/dL)
* Probable diabetes: HbA1c >6.0

Contraindication to a component of the Polypill

Contraindications to aspirin

* Previous history of allergy to aspirin
* History of peptic ulcer bleeding in whole life or endoscopic evidence of peptic ulcer within the past 3 months

Contraindications to statins

* Liver failure Contraindications to further blood pressure lowering
* Systolic blood pressure ≤90 mm Hg or diastolic blood pressure ≤70 mm Hg
* Symptomatic postural hypotension
* Difference between mean seated BP and standing BP greater than 20 mm Hg

Contraindications to thiazide

* Uric acid >8 for men and uric acid >6 for women / gout (~10%)
* Creatinine >1.2 mg/dl

Other predominant medical problem that may limit compliance with study treatment including:

* History of alcohol abuse: more than 60cc for women and more than 80cc for men
* History of drug abuse: IV drug abuser or eating or smoking more than 4 times a week
* Limiting psychiatric illness (eg: mania, schizophrenia, severe depression, psychosis or dementia)
* Limiting physical disability sufficient to prevent subject from walking
* Other life-threatening condition such as cancer

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 475 (Actual)
Dates: Start 2006-11; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reza Malekzadeh, M.D., Study Chair — Tehran University of Medical Sciences; Fatemeh Malekzadeh, M.D., Principal Investigator — Tehran University of Medical Sciences; Mansoor Rastegarpanah, Ph.D., Principal Investigator — Tehran University of Medical Sciences; Kar K Cheng, PhD, Study Chair — University of Birmingham; Tom P Marshall, PhD, Principal Investigator — University of Birmingham; Akram Pourshams, PhD, Study Director — Tehran University of Medical Sciences
Locations (1):
- Kalaleh Heart Study Center, Kalāleh, Golestan Province, Iran

REFERENCES:
- [Background] Rastegarpanah M, Malekzadeh F, Thomas GN, Mohagheghi A, Cheng KK, Marshall T. A new horizon in primary prevention of cardiovascular disease, can we prevent heart attack by "heart polypill"? Arch Iran Med. 2008 May;11(3):306-13. No abstract available. PMID 18426322

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between July 2006 and January 2007, 1,733 subjects attended the Kalaleh heart clinic. Of those assessed 872 were included in the run-in phase of the study. Of these 475 were randomized.
Pre-assignment Details: 872 subjects entered the run in phase, 258 were excluded. Most exclusions were due to laboratory test results.
  614 completed the run-in phase of the study, 65 were excluded. Most were excluded because they did not attend the clinic.
  Of 549 subjects remaining, 74 were not randomized.
  475 subjects who were randomized.
Groups:
- Polypill: Polypill (Atorvastatin 20 mg, Asprin 81 mg, Enalapril 2.5 mg, Hydrochlorothiazide 12.5 mg)
- Control: Identical placebo tablet
Period: Overall Study
Arm/Group | Polypill | Control
Started | 241 | 234
One Month | 204 | 212
Four Months | 187 | 200
Eight Months | 178 | 194
Completed | 165 | 183
Not Completed | 76 | 51
Not completed — Did not attend study clinic | 39 | 30
Not completed — Refused blood test | 5 | 1
Not completed — Patient discontinued study drug | 22 | 15
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 8 | 4
Not completed — Cardiovascular event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Polypill | Control | Total
Number analyzed (Participants) | 241 | 234 | 475
Age Continuous [Mean (Standard Deviation); unit: Years] | 59.0 (6.5) | 59.1 (7.3) | 59.0 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 67 | 158
  Male | 150 | 167 | 317
Region of Enrollment [Number; unit: participants]
  Iran, Islamic Republic of | 241 | 234 | 475
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] — Mean of two seated blood presures
  mm Hg | 78.4 (10.4) | 81.2 (9.7) | 79.8 (10.1)
LDL cholesterol [Mean (Standard Deviation); unit: mg/dL] — Serum LDL cholesterol levels
  mg/dL | 116.7 (25.8) | 116.6 (24.8) | 116.6 (25.2)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] — Mean of two seated systolic blood pressures
  mm Hg | 124.8 (17.3) | 130.3 (17.4) | 127.5 (17.5)

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure
Description: Systolic blood pressure. Mean of two seated measurements.
Time Frame: One year
Population: Intention to treat Results shown here are based on 12 month observation. Analysis for final paper will be last observation carried forward
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Polypill | Control
Number analyzed (Participants) | 165 | 183
mm Hg | 121.7 (16.8) | 129.7 (18.3)

2. Secondary Outcome: Diastolic Blood Pressure
Description: Mean of two seated diastolic blood pressures
Time Frame: One year
Population: Analysis by intention to treat. Results shown here are based on 12 month observation. Analysis for final paper will be last observation carried forward.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Polypill | Control
Number analyzed (Participants) | 165 | 183
mm Hg | 77.6 (10.6) | 81.3 (11.1)

3. Secondary Outcome: LDL Cholesterol
Description: Serum LDL cholesterol
Time Frame: One year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Polypill | Control
Number analyzed (Participants) | 160 | 175
mg/dL | 87.8 (26.7) | 112.0 (26.8)

ADVERSE EVENTS:
Arm/Group | Polypill | Control
Serious Adverse Events (participants affected / at risk) | 0 | 1
Other Adverse Events (participants affected / at risk) | 2 | 0
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Polypill | Control
Cardiovascular event (Cardiac disorders) | 0/241 (0) | 1/234 (1)
OTHER ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Polypill | Control
Cough (Respiratory, thoracic and mediastinal disorders) | 2/241 (2) | 0/234 (0)

LIMITATIONS AND CAVEATS:
Incomplete follow up Because of differences in systolic blood pressure at baseline, final analysis will take account of baseline differences

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No